CLINICAL TRIAL: NCT06527677
Title: Phase 1, Open-Label, Non-Randomized, Single-Center, Single-Dose Study to Assess the Pharmacokinetics & Safety of ANT3310 Combined With Meropenem Administered as a Single Intravenous Infusion to Adult Subjects With Renal Function Impairment
Brief Title: Assessment of the Pharmacokinetics and Safety of ANT3310 Combined With Meropenem in Renally Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antabio (Industry)
Collaborators: Clinical Research Center Kiel GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ANT3310-1002
Record Dates: First submitted 2024-07-08; First posted 2024-07-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ANT3310 and Meropenem (Experimental): Participants with mild, moderate, or severe renal function impairment (Panel A, B, and D) and participants with normal renal function (Panel C and F) will receive 1 single dose of a combination of ANT3310 and meropenem.
  Participants with End Stage Renal Disease (Panel E) will receive 2 times a single dose of a combination of ANT3310 and meropenem: one single dose during dialysis-free interval ("off- dialysis") and one single dose on the day of dialysis ("on-dialysis"). The same dose will be given in both periods with a washout interval of at least 7 days between administrations.
  Interventions: Drug: ANT3310; Drug: Meropenem

INTERVENTIONS:
Drug: ANT3310 — ANT3310 will be administered as a single intravenous infusion over 3 hours at a constant rate.
Drug: Meropenem — meropenem will be administered as a single intravenous infusion over 3 hours at a constant rate.

SUMMARY:
This is an open-label, non-randomized, single-center, single i.v. dose Phase 1 trial to evaluate the pharmacokinetics and safety of a combination of ANT3310 and meropenem in participants with different degrees of renal function impairment, including participants with End-Stage Renal Disease (ESRD), compared with matching control participants with normal renal function.

DETAILED DESCRIPTION:
The participants will receive 1 single dose of the combination of ANT3310 and meropenem (2 times a single dose in participants with ESRD).

ELIGIBILITY:
Main Inclusion Criteria:

* Participant must be 18 to 80 years of age (both inclusive) at the time of signing the informed consent.
* BMI within the range of 18.0 to 36.0 kg/m2 (both inclusive) with a body weight ≥ 50 kg.
* Contraceptive use by women or men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent in compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Ability to cooperate with the investigator and to comply with the requirements of the trial.
* Sufficient venous access for i.v. infusion and PK samplings.
* For participants with renal function impairment: Individualized eGFR <90 mL/min at screening, estimated according to the individualized CKD-EPI equation and stable renal function.
* For participants with ESRD requiring dialysis: Chronic intermittent hemodialysis for ≥3 months prior to dosing.
* For participants with normal renal function: Individualized eGFR ≥90 mL/min at screening, estimated based on serum creatinine measured within 10 days prior to Day -1 according to the CKD-EPI equation.

Main Exclusion Criteria:

* Febrile illness within 1 week before admission to the study center.
* Known hypersensitivity to meropenem and or ANT3310 or any of the excipients of the infusion solution.
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies requiring intranasal or systemic corticosteroids during any time of the year or history of any anaphylactic reaction.
* Medical disorder, condition, or history of such that would - in the opinion of the investigator - compromise the participant's ability to participate in this study.
* History of epilepsy (or known seizure disorder), brain lesions or other significant neurological disorders.
* Known history of clinically significant hypersensitivity or urticaria, or severe allergic reaction to β-lactam antibiotics (e.g., penicillin, cephalosporin, carbapenem, or monobactam).
* History of Gilbert syndrome.
* History of any severe antibiotic-associated superinfections like Clostridium difficile colitis and/or frequent fungal vaginal infections.
* Therapies (e.g., physiotherapy, acupuncture, etc.) within 1 week before study drug administration.
* Positive results for HBsAg, anti-HCV, HIV antibodies (anti-HIV 1+2).
* For participants with impaired renal function: Acute renal failure or active renal infections, Clinically significant impaired hepatic function, Severe infection or any clinically significant illness within 4 weeks before dosing, Impairment of any other major organ system other than the kidney except underlying disease, Diagnosed malignancy during the past 5 years except completely resected basal cell cancer of the skin, Any kidney transplant during the last 10 years, any other organ transplant during the past 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentrations (Cmax) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Area under the curve from 0 to infinity (AUC0-inf) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Time from dosing to maximum observed concentration (tmax) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Apparent terminal elimination half-life (t1/2λz) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Area under the curve from time 0 to time of last measurable concentration (AUC0-last) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Area under the curve from time 0 to 48h (AUC0-48h) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Percentage of AUC0-inf obtained by extrapolation (AUCext) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Total body clearance (CL) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Non-renal clearance (CLNonR) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma and urine.
Apparent volume of distribution during the terminal phase after administration (Vz) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Mean residence time (MRT) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in plasma.
Amount of ANT3310 and Meropenem that is eliminated in urine from 0 to infinity (Ae0-inf) after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in urine.
Renal clearance (CLR) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in urine.
Fraction of dose recovered in urine (fe) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in urine.
Amount of ANT3310 and Meropenem that is eliminated in urine from 0 to 48h (Ae0-48h) after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in urine.
Fraction of dose recovered in urine from 0 to 48 hours (fe0-48h) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in urine.
Renal clearance from 0 to 48 hours (CLR[0-48h]) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem | From pre-dose to Day 3
  Pharmacokinetic parameter of ANT3310 and Meropenem in urine.
Dialysis clearance (CLD) of ANT3310 and Meropenem after a single i.v. infusion of the combination ANT3310-Meropenem in dialysed subjects | during dialysis
  Pharmacokinetic parameter of ANT3310 and Meropenem in dialysate and plasma.

SECONDARY OUTCOMES:
Number and severity of treatment-emergent adverse event (TEAE) to evaluate the safety and tolerability of ANT3310 and meropenem after a single i.v. infusion of a combination of ANT3310 and meropenem. | 0 hours to Day 9
  Percentage of participants experiencing ≥ one treatment-emergent adverse event (TEAE) by seriousness, intensity, and relatedness from baseline to end of study (EoS) or early withdrawal.
Number of participants who discontinue due to a TEAE. | 0 hours to Day 9
  Percentage of participants who discontinue due to a TEAE.
Number of participants who meet the clinically significant abnormal criteria for safety laboratory tests at least once after start of dosing. | 0 hours to Day 9
  Percentage of participants who meet the clinically significant abnormal criteria for safety laboratory tests at least once after start of dosing.
Number of participants meeting the clinically significant abnormal criteria for vital signs measurements at least once after start of dosing. | 0 hours to Day 9
  Percentage of participants meeting the clinically significant abnormal criteria for vital signs (blood pressure, pulse rate, respiratory rate, and body temperature) measurements at least once after start of dosing.
Number of participants who meet the clinically significant abnormal criteria for ECG (Electrocardiogram) parameters. | Day-1 to Day 9
  Percentage of participants who meet the clinically significant abnormal criteria for ECG parameters.
Number of infusion site reactions to assess local venous tolerability | From pre-dose on Day 1 to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Christian Zwingelstein, PharmD, Study Director — Antabio
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No